CLINICAL TRIAL: NCT02363764
Title: The Challenge of Obtaining Qualitative Bacterial Cultures in Non-expectorating Cystic Fibrosis Patients
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Hanneke Eyns, Physiotherapist, Universitair Ziekenhuis Brussel
Other Study IDs: B.U.N. 143201422976
Record Dates: First submitted 2015-01-30; First posted 2015-02-16 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Cystic Fibrosis
Keywords: respiratory sampling
MeSH Terms: conditions — Cystic Fibrosis | interventions — Bronchoalveolar Lavage; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Expectorating CF patients: (=able to expectorate sputum spontaneously)
  1. Nasal swab
  2. Cough swab
  3. Spontaneous expectorated sputum
  4. Questionnaire
  Interventions: Procedure: Nasal swab; Procedure: Cough swab; Procedure: Spontaneous expectorated sputum; Other: Questionnaire
- Non-expectorating CF patients: (=unable to expectorate sputum spontaneously)
  1. Nasal swab
  2. Cough swab
  3. Induced sputum after inhalation of hypertonic saline (NaCl 6%)
  4. Questionnaire
  Interventions: Procedure: Nasal swab; Procedure: Cough swab; Procedure: Induced sputum; Other: Questionnaire
- Bronchoscopy CF patients: (=undergoing clinically indicated bronchoscopy)
  1. Nasal swab
  2. Cough swab
  3. Induced sputum after inhalation of hypertonic saline (NaCl 6%)
  4. Bronchoalveolar lavage (BAL)
  Interventions: Procedure: Nasal swab; Procedure: Cough swab; Procedure: Induced sputum; Procedure: Bronchoalveolar lavage

INTERVENTIONS:
Procedure: Nasal swab — Will be obtained by the physiotherapist in:
  * Expectorating CF patients
  * Non-expectorating CF patients
  * Bronchoscopy CF patients
Procedure: Cough swab — Will be obtained by the physiotherapist in:
  * Expectorating CF patients
  * Non-expectorating CF patients
  * Bronchoscopy CF patients
Procedure: Spontaneous expectorated sputum — Will be obtained by the physiotherapist in:
  - Expectorating CF patients
  Groups: Expectorating CF patients
Procedure: Induced sputum — Will be obtained by the physiotherapist in:
  * Non-expectorating CF patients
  * Bronchoscopy CF patients
  Groups: Bronchoscopy CF patients; Non-expectorating CF patients
Procedure: Bronchoalveolar lavage — Will be obtained by the pulmonologist in:
  - Bronchoscopy CF patients
  Groups: Bronchoscopy CF patients
Other: Questionnaire — Completing questionnaire on acceptability of different sampling methods by patients >6 years of age
  Groups: Expectorating CF patients; Non-expectorating CF patients

SUMMARY:
Accurate identification of lower respiratory tract pathogens is standard of care in the management of CF patients and it is therefore recommended to perform regular bacterial cultures, at least once a year, but some even recommend monthly cultures. This can be done through different methods, of which sputum and bronchoalveolar lavage (BAL) are the gold standard. However, BAL is an invasive method, not designated to repeat monthly. Therefore, the diagnosis of lower respiratory tract infections can be challenging in the non-expectorating CF patient. Other methods, such as induced sputum (IS), cough swabs and nasal swabs, have been developed to obtain bacterial cultures in these patients. Studies have investigated the reliability of these different sampling methods, however, with controversial conclusions.

DETAILED DESCRIPTION:
I. Protocol design:

The current protocol is designed to compare:

* Group 1: nasal swab, cough swab and spontaneous expectorated sputum in expectorating CF patients
* Group 2: nasal swab, cough swab and induced sputum in non-expectorating CF patients
* Group 3: nasal swab, cough swab, induced sputum and BAL in both expectorating and non-expectorating CF patients requiring clinically indicated bronchoscopy

II. Flow chart:

1. Nasal swab obtained by the physiotherapyst (PT)
2. Patient rinses his mouth with water, followed by autogenic drainage
3. Cough swab obtained by the PT
4. Obtainment of 3rd (4th) sample:

   * Group 1: Sputum sample voluntary expectorated by the patient
   * Group 2 and 3: Induced sputum sample --> voluntary coughed up and expectorated by the patient after inhalation of 4ml of HS OR
   * Group 3: BAL -->obtained by the pulmonologist during bronchoscopy
5. Filling out questionnaire on acceptability of the different sampling methods by patients >6 years of age (not in Group 3)

III. Analysis of the samples:

(Induced) Sputum samples, cough and nasal swabs are aseptically collected in the appropriate disposable and are immediately sent to the Laboratory for Microbiology and Infection Control of the Universitair Ziekenhuis Brussel, where analyses are carried out within 24h post-sampling.

These analyses include:

* Culture and identification of respiratory pathogens on selective and non-selective media
* Each type of colony will be identified by MALDI-TOF mass spectrometry, completed by other identification tests if needed
* When appropriate, susceptibility tests will be performed on the isolated bacteria

IV. Statistical analysis:

* Determination of sensitivity, specificity, positive predicted value, negative predicted value of the different sampling methods
* Preference for one method over another: crosstabs, Chi-square test
* Pain experienced with any method (Yes/No): Student's t-test
* VAS-scale pain per method: ANOVA

ELIGIBILITY:
Inclusion Criteria:

* Both expectorating and non-expectorating CF patients with confirmed diagnosis (sweat test / genotyping)
* All ages
* Attending the UZ Brussel CF Clinic
* Written informed consent from each participant and/or his parents or legal guardian

Exclusion Criteria:

* CF patients who underwent lung transplantation
* Denial of participation to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive and negative predicted value | 2 years
  Sensitivity, specificity, positive and negative predicted value of different sampling methods

SECONDARY OUTCOMES:
Preference of method | Questionnaire: day of sampling, Analysis: 2 years
  If no differences are observed between sampling methods, which method would be preferred by the patient?
Pain experienced with any method | Questionnaire: day of sampling, Analysis: 2 years
  Is there any pain experienced? If so, how much? --> VAS

CONTACTS AND LOCATIONS:
Overall Officials: Anne Malfroot, MD, PhD, Study Director — Universitair Ziekenhuis Brussel - Cystic Fibrosis Clinic

IPD SHARING:
Plan to Share IPD: No
All data will be analysed and shared as an original article, individual data will only be available upon motivated request